CLINICAL TRIAL: NCT00912340
Title: Phase II Trial of EVEROLIMUS ± Trastuzumab in Hormone-Refractory Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Genentech, Inc. (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Elisavet Paplomata, Principal Investigator, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012495; WCI1524-08 (Other: Other)
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Trastuzumab (Experimental): Patients receive trastuzumab IV over 30 minutes once every 3 weeks and continue to receive their most recent hormone therapy. Patients achieving disease progression receive everolimus PO daily in combination with trastuzumab and hormone therapy.
  Interventions: Biological: Trastuzumab
- Everolimus (Experimental): Patients receive everolimus PO daily and continue their most recent hormone therapy. Patients achieving disease progression receive trastuzumab IV over 30-90 minutes once every 3 weeks in combination with everolimus and hormone therapy.
  Interventions: Drug: Everolimus
- Trastuzumab and everolimus (ARM REMOVED) (Experimental): Patients receive trastuzumab IV over 30 minutes once every 3 weeks and everolimus PO daily while continuing to receive their most recent hormone therapy.
  Interventions: Drug: Everolimus; Biological: Trastuzumab

INTERVENTIONS:
Drug: Everolimus
  Other Names: Afinitor; RAD001
  Arms: Everolimus; Trastuzumab and everolimus (ARM REMOVED)
Biological: Trastuzumab
  Other Names: Herceptin
  Arms: Trastuzumab; Trastuzumab and everolimus (ARM REMOVED)

SUMMARY:
This phase II trial studies how well everolimus with or without trastuzumab works in treating patients with breast cancer that has not responded to hormone therapy and has spread from where it started to other places in the body. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as trastuzumab, may interfere with the ability of tumor cells to grow and spread. Giving everolimus and adding trastuzumab at the time of disease progression may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common type of invasive cancer in women, with more than 1 million cases and almost 600,000 deaths occurring worldwide annually. Breast cancer that has spread to other parts of the body (metastasized) is usually not curable. Patients with a type of metastatic breast cancer that has hormone receptors on the surface of the cancer cells are usually treated with the drug tamoxifen, which interferes with the function of these hormone receptors. However, the average survival time for these patients remains at around 36 months.

In patients who no longer respond to tamoxifen (hormone-refractory breast cancer), the cancer drug trastuzumab (Herceptin), which acts on a protein called human epidermal growth factor receptor 2 (HER2), may have some activity. In addition, studies suggest that the drug everolimus, which acts on a pathway within cancer cells that is important for growth of the tumor, may make the cancer cells more sensitive to treatment with trastuzumab. Thus, the two drugs may act together to increase their anti-cancer potential.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study based on the following criteria:

* Hormone-refractory metastatic breast cancer defined as disease progression within 6 months from starting most recent hormonal therapy
* At least one line of endocrine therapy in the metastatic setting
* Candidate for hormonal therapy (ER and/or progestin receptor [PR]-positive at primary diagnosis and at metastatic diagnosis where tissue is available)
* HER2/neu-negative breast cancer by standard criteria (immunohistochemistry [IHC] < 3+ or fluorescence in situ hybridization [FISH]-negative if IHC 3+) at primary diagnosis
* Must have a biopsy in the metastatic setting with HER2 expression of 1+ or 2+ by IHC
* If biopsy of metastatic lesion is performed prior to study entry, HER2 expression by IHC must be 1+ or 2+
* Histologically confirmed, measurable or evaluable disease; if disease is measurable, Response Evaluation Criteria In Solid Tumors (RECIST) criteria should be used
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate bone marrow function as indicated by the following:

  * Absolute neutrophil count (ANC) > 1500/µL
  * Platelets ≥ 100,000/µL
  * Hemoglobin > 10 g/dL
* Adequate renal function, as indicated by creatinine ≤ 1.5x upper limit of normal (ULN)
* Adequate liver function, as indicated by bilirubin ≤ 1.5x ULN
* International normalized ratio (INR) ≤ 1.3 (or ≤ 3 on anticoagulants)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2x ULN unless related to primary disease
* Signed informed consent
* Adequate birth control
* Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.

Exclusion Criteria:

Patients will be excluded from the study based on the following criteria:

* Prior treatment with trastuzumab or other HER2-directed therapies or with an mammalian target of rapamycin (mTOR) inhibitor within 12 months of study entry (when cancer was not definitely hormone refractory)
* HER2 0 or 3+ by IHC on pre-treatment biopsy of metastatic lesion (if performed)
* Active infection
* Uncontrolled central nervous system metastases
* Life-threatening, visceral metastases
* Pregnant or lactating women
* Prior chemotherapy within the last 4 weeks
* Prior radiation therapy within the last 4 weeks; prior radiation therapy to indicator lesion (unless objective disease recurrence or progression within the radiation portal has been documented since completion of radiation)
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* History of significant cardiac disease, cardiac risk factors or uncontrolled arrhythmias
* Ejection fraction < 50% or below the lower limit of the institutional normal range, whichever is lower
* Hypersensitivity to trial medications
* Emotional limitations
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent
* Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods. If barrier contraceptives are being used, these must be continued throughout the trial by both sexes. Hormonal contraceptives are not acceptable as a sole method of contraception. (Women of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to administration of everolimus)
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus)
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest
* Taking any of the following agents:

  * Chronic treatment with systemic steroids or another immunosuppressive agent
  * Live vaccines
  * Drugs or substances known to be inhibitors or inducers of the isoenzyme cytochrome P450, family 3, subfamily A (CYP3A)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisavet Paplomata, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (4):
- United States (4):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at Winship Cancer Institute of Emory University, Emory University Hospital Midtown, and Robert H. Lurie Comprehensive Cancer Center of Northwestern University.
Pre-assignment Details: 70 participants were enrolled. Nine were found to be ineligible. Three declined to participate and were not treated.
Period: Overall Study
Arm/Group | Trastuzumab | Everolimus | Trastuzumab and Everolimus (ARM REMOVED)
Started | 24 | 30 | 4
Completed | 22 | 26 | 0
Not Completed | 2 | 4 | 4
Not completed — Adverse Event | 2 | 4 | 0
Not completed — Protocol revised to remove arm | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab | Everolimus | Trastuzumab and Everolimus (ARM REMOVED) | Total
Number analyzed (Participants) | 24 | 30 | 4 | 58
Age, Customized [Count of Participants; unit: Participants]
  Age range 30-39 | 2 | 0 | 0 | 2
  Age range 40-49 | 2 | 5 | 0 | 7
  Age range 50-59 | 9 | 8 | 0 | 17
  Age range 60-69 | 4 | 9 | 4 | 17
  Age range 70-79 | 7 | 7 | 0 | 14
  Age range 81-89 | 0 | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 4 | 57
  Male | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 23 | 26 | 4 | 53
  Unknown or Not Reported | 1 | 3 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 3 | 1 | 13
  White | 15 | 24 | 2 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 30 | 4 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Until First Progression
Description: Median PFS will be calculated based on time to first progression or death.
Time Frame: Every 3 to 4 weeks after study start, until progression or death, assessed up to 5 years
Population: Four patients were treated with both trastuzumab & everolimus up front. These patients were not included in the data analysis because this arm was later discontinued.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab | Everolimus | Trastuzumab and Everolimus (ARM REMOVED)
Number analyzed (Participants) | 24 | 30 | 0
months | 2.0 [1.6 to 4.1] | 5.7 [3.9 to 8.9] |

2. Secondary Outcome: Progression-free Survival (PFS) in Patients Who Crossed Over
Description: Median PFS will be calculated based on time to first progression or death.
Time Frame: Every 3 to 4 weeks after study start, until progression or death, assessed up to 5 years
Population: Among 48 patients with disease progression, everolimus was added to 16 patients treated by trastuzumab, and trastuzumab was added to 12 patients treated by everolimus.
  Four patients were treated with both trastuzumab & everolimus up front. These patients were not included in the data analysis because this arm was later discontinued.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab | Everolimus | Trastuzumab and Everolimus (ARM REMOVED)
Number analyzed (Participants) | 16 | 12 | 0
months | 6.3 [2.6 to 10.5] | 3.1 [1.8 to 6.7] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study assessed up to 5 years. Patients were evaluated in the clinic every 3 weeks and then after a protocol amendment, they were evaluated every 4 weeks if only receiving everolimus plus endocrine therapy and not trastuzumab. Scans were done at 6 weeks from the start of treatment and then every 12 weeks.
Groups:
- Trastuzumab: Patients receive 10 mg everolimus PO daily and continue to receive their most recent hormone therapy. Patients achieving disease progression receive 8 mg/kg trastuzumab IV over 30-90 minutes once every 3 weeks in combination with everolimus and hormone therapy.
Arm/Group | Trastuzumab | Everolimus | Trastuzumab and Everolimus (ARM REMOVED)
All-Cause Mortality (participants affected / at risk) | 9/24 | 8/30 | 3/4
Serious Adverse Events (participants affected / at risk) | 1/24 | 6/30 | 0/4
Other Adverse Events (participants affected / at risk) | 0/24 | 12/30 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=24) | Everolimus (N=30) | Trastuzumab and Everolimus (ARM REMOVED) (N=4)
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0
Other cardiac disorder (Cardiac disorders) | 0 | 1 | 0
Ejection fraction decrease (Cardiac disorders) | 0 | 1 | 0
Hypertension (General disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Salivary gland infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab (N=24) | Everolimus (N=30) | Trastuzumab and Everolimus (ARM REMOVED) (N=4)
Aspartate aminotransferase (AST) increased (Investigations) | 0 | 1 | 0
Alanine aminotransferase (ALT) increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 2 | 0
Edema limbs (General disorders) | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decreased ejection fraction (Investigations) | 0 | 2 | 0
Angioedema (General disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
Since the initial study design would not allow evaluation of everolimus alone, in 2010, the protocol was amended so that patients were randomized to trastuzumab or everolimus. In 2014, the protocol was amended to close the trastuzumab arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Trial design changed (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT00912340/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Former trial design (2014-03-07): https://cdn.clinicaltrials.gov/large-docs/40/NCT00912340/Prot_SAP_001.pdf